CLINICAL TRIAL: NCT02971449
Title: Using mHealth Tools to Deliver Integrated Community Case Management (ICCM) to Village Health Team (VHT) Volunteers in Uganda.
Brief Title: Using mHealth Tools to Deliver Integrated Community Case Management (ICCM) to Village Health Team (VHT) Volunteers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Omni Med (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BMAChartiableGrant2016
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Community Health Services; Telemedicine
Keywords: Village Healthcare Team; mHealth; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tablets only (Experimental): 100 VHTs will receive Amazon Fire Tablets with pre-loaded instructional videos; this is the intervention arm since this involves introduction of a new technology to this realm
  Interventions: Device: Amazon Fire Tablet
- ICCM traditional training (Active Comparator): 100 VHTs will receive traditional 1 day 'in-person' training as an active comparator intervention, but participants in this arm will not receive any tablets
  Interventions: Other: ICCM Traditional Trainins

INTERVENTIONS:
Device: Amazon Fire Tablet — A generic amazon fire tablet with pre-loaded instructional videos
  Arms: Tablets only
Other: ICCM Traditional Trainins — Standard, Didactic VHT Training intervention as an active comparator
  Arms: ICCM traditional training

SUMMARY:
This study compares the traditional, didactic method of training Ugandan community health workers with training using tablets in pneumonia management, a common, life-threatening illness in children in rural areas.

DETAILED DESCRIPTION:
Current ICCM (Integrated Community Case Management) training in Uganda involves CHWs physically attending a five-day workshop, which is both expensive, time consuming and requires trainer's to be physically present to deliver training materials. The investigators hypothesize that use of a low-cost android tablet, with pre-loaded instructional educational videos will improve the baseline knowledge and retention of knowledge of CHWs as well as lower the direct and indirect costs of ICCM training.

The investigators will conduct a randomized controlled trial in two sub-counties in Mukono district among CHWs to test these two hypotheses. In this study, the investigators will focus solely on the pneumonia component of ICCM training, instead of testing the full week-long training course including malaria, pneumonia, and diarrhea. (The investigators plan a later trial encompassing the entire week-long training vs the same uploaded into the tablets.) The investigators will enroll 200 CHWs in the study, with 100 in a control group who will receive a one day in-person training session focusing on pneumonia, similar to traditional ICCM training and 100 in an intervention group who will receive tablets with instructional training videos. The investigators will administer a written test prior to the training in both groups, then administer the same written test one week later. Additionally, the investigators will test both groups with clinical case scenarios that give these community health workers realistic clinical cases and challenge them to diagnose pneumonia, state whether patient should be treated in the home or brought to hospital, and how to initiate and complete management if patients are to be referred or kept home, respectively. The sample sizes will enable the investigators carry out independent t-tests and a paired two-sample t-test to determine the significance of pre- and post-test scores for the control and intervention groups. If training delivered via low-cost android tablets proves to be both effective and acceptable, this option may represent a viable, scalable and cost-effective alternative to the traditional training model used throughout Uganda.

Furthermore, the MoH could institute an incentive policy that allows tablets to be distributed and retained by health workers provided that they maintain a quarterly flow of information back to the MoH regarding home visits, patients referred, or other community actions. Should the learning and cost efficacy prove viable, the investigators can envision tablets throughout Mukono District, allowing the more direct transfer of information, disease patterns, index cases of pathogens like Ebola, tracking of data for the Ministry, regular dissemination of training materials, and opportunities for CHWs gain employment in the health sector.

ELIGIBILITY:
Inclusion Criteria:

* Must be a registered VHT working in the study areas in Uganda;
* Must express a commitment to aim to complete the duration of the study;
* Willingness to be randomised to the control or intervention group.

Exclusion Criteria:

- Unregistered VHTs

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Is VHT knowledge retention comparable or superior when comparing the use of tablets with standard Ugandan ICCM training methods in the recognition and management of pneumonia in children by Ugandan VHTs? | 2 months
  There will be 2 arms of the study to see if pre-loaded instructional videos on a low cost android tablet are either superior to or comparable to standard training methods in the training of VHTs in Mukono, Uganda in terms of recognition, prevention and management of pneumonia in children under 5 years old in line with ICCM guidelines. One group will receive normal ICCM training by attending the standard, didactic ICCM training workshop held in the community. The second, Interventional arm will utilize Ministry approved training videos pre-loaded into low cost android tablets. The overall aim of the study is to assess whether or not the tablets can replace the current time-consuming and expensive methods used throughout Uganda.

SECONDARY OUTCOMES:
Cost efficacy of the Tablet Approach to ICCM Training | 2 months
  We will perform detailed cost analysis for both arms of this trial. Generally, it is expensive to bring a group of VHTs together for trainings, with costs including transport, food, instructors, petrol, and materials. By contrast, getting tablets out to VHTs with simple user instructions allows learning to happen at home, and repeatedly by watching the videos over and over again.

CONTACTS AND LOCATIONS:
Overall Officials: Edward J O'Neil Jr, MD, Principal Investigator — Omni Med; James O'Donovan, MD, Principal Investigator — Omni Med
Locations (2):
- Omni Med, Newton, Massachusetts, United States
- Omni Med, Kisoga, Mukono, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Donovan J, Kabali K, Taylor C, Chukhina M, Kading JC, Fuld J, O'Neil E. The use of low-cost Android tablets to train community health workers in Mukono, Uganda, in the recognition, treatment and prevention of pneumonia in children under five: a pilot randomised controlled trial. Hum Resour Health. 2018 Sep 19;16(1):49. doi: 10.1186/s12960-018-0315-7. PMID 30231894